CLINICAL TRIAL: NCT01860872
Title: Study of Cardiac MRI to Assess Pulmonary Perfusion and Pulmonary Hemodynamics in Patients With Cystic Fibrosis Study (Pilot 3)
Brief Title: Comparing Chest Images From MRI to CT in Patients With Cystic Fibrosis (CF)
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CIN001-CF MRI; 1R01HL116226-01 (NIH)
Record Dates: First submitted 2013-05-15; First posted 2013-05-23 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2018-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Pulmonary perfusion; Inflammatory markers; MRI; CT of chest; Lung Clearance Index
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CF Group: Cystic Fibrosis group with MRI and CT of chest
- Control group: Non-CF controls will have MRI and no CT of chest
- Combined Group: MRI Quality & Image Relatedness

SUMMARY:
The purpose of this research is to learn more about the heart and blood vessels in the lungs of people with cystic fibrosis (CF). This study will include approximately 36 children and adults with CF and 12 children and adults without CF. The study will involve one magnetic resonance imaging (MRI) . The research also includes blood samples to look at inflammation and lung tests called spirometry and Lung Clearance Index (LCI) determined by Multiple Breath Washout test.

For the CF subjects, enrollment will be timed to coincide with routine scheduled computerized tomography (CT) or the CF subject may choose to have a CT for research purposes. The MRI will be compared to CT images of the lungs. The goal is to develop better imaging that does not use radiation.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF), the most common inherited disease in Caucasians, is characterized by chronic pulmonary inflammation and progressive loss of gas exchange units that eventually results in respiratory failure. There is strong evidence that in CF abnormally low vascular perfusion carries a high risk of death independent from the presence of pulmonary hypertension. However, the evolution of pulmonary vascular disease in CF and how it might contribute to the rate of decline in lung function is not known. Knowledge remains limited to the results of old observational studies which concluded that the major causes of pulmonary vascular remodeling and hypertension in CF are hypoxic respiratory failure and destruction of lung tissue. Recent data obtained by state-of-the-art Magnetic Resonance Imaging (MRI) of the pulmonary circulation, challenges the existing paradigm. Studies demonstrate that in the absence of hypoxia, significant changes in pulmonary perfusion and in surrogate measures of vascular resistance as well as in collateral blood flow begin early in the course of CF. The newly developed therapeutics in the last decade which altered dramatically the course of patients suffering from pulmonary vascular disease provide opportunities to understand the role of pulmonary vasculature in CF lung disease.

This pilot study (Pilot 3) will assess the relationships between pulmonary perfusion, serum markers of pulmonary inflammation and vascular remodeling, and hemodynamic measures consistent with pulmonary hypertension. This study will establish MRI as a readily obtainable modality to be used in the CF population to obtain measurements of pulmonary perfusion; pulmonary arterial hemodynamic, dimension, and flow measures; and ventricular mass and function measures.

The primary goal of this study is to improve the understanding of pulmonary vascular disease in CF by examining pulmonary perfusion abnormalities and their association with markers of pulmonary inflammation and pulmonary vascular remodeling, the severity of obstructive airways disease, and pulmonary hemodynamic abnormalities in CF.

This study will include a single MRI of the pulmonary circulation on about 36 pediatric and adult patients with CF and about 12 non-CF controls. UTE (Ultrashort Echo Time) MRI will be performed without contrast. CF patients who are scheduled for clinical chest CT will be enrolled and the scheduling of the MRI will be coordinated with the clinical CT. CF subjects may also choose to enroll independent of clinical CT and choose to have a CT for research purposes only. Other study procedures include blood specimen for serum biomarkers and lung tests called spirometry and Lung Clearance Index (LCI) determined by Multiple Breath Washout test. Blood specimens will be analyzed for a panel of inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 and older
* Diagnosis of cystic fibrosis confirmed by a prior sweat chloride evaluation of > 60 mmol/liter or by two identified CF mutations on genetic analysis; or no CF for controls
* Able to perform acceptable and repeatable spirometry per American Thoracic Society/European Respiratory Society (ATS/ERS) joint consensus criteria.
* If CF, have valid spirometry data for at least 3 years
* If under the age of 18, the patient must assent to participation in the study, and the patient's parent or guardian must be able to give written informed consent and comply with the requirements of the study protocol
* If 18 years of age or older, the patient must be able to give written informed consent and comply with the requirements of the study protocol
* Negative serum pregnancy test (for women of child bearing age)
* Able to tolerate MRI without sedation

Exclusion Criteria:

* Pregnancy (a negative serum pregnancy will be performed for all women of childbearing potential within 7 days of imaging) or lactation
* Subjects with a history of renal
* Subjects with a history of hypersensitivity to gadolinium (Magnevist)
* Contraindications specific to MRI including a history of claustrophobia, cardiac pacemaker, or other non-MRI compatible surgical implants (This includes neuro-stimulators containing electrical circuitry, or which generate electrical signals and/or have moving metal parts, and metal orthopedic pins or plates. The research coordinator and/or the MRI technologist will screen all patients using the standard checklist of medical history and safety questions used by the Radiology Department in routine clinical scans.)
* Inability to comply with study procedures

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cystic Fibrosis and Non-CF Controls
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary MRI and CT | Baseline (MRI and CT acquisition)
  Assess perfusion in each pulmonary segment. Segmental perfusion will be scored on a continuous scale (0=normal, 1=mild abnormality, 2=moderate abnormality, 3=severe abnormality) for each of the 18 lobar segments.

CONTACTS AND LOCATIONS:
Overall Officials: John Clancy, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States